CLINICAL TRIAL: NCT01773707
Title: CTLA4-Ig (Abatacept)for Prevention of Abnormal Glucose Tolerance and Diabetes in Relatives At -Risk for Type 1 Diabetes
Brief Title: CTLA4-Ig (Abatacept)for Prevention of Abnormal Glucose Tolerance and Diabetes in Relatives At -Risk for Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: Abatacept (IND); UC4DK106993 (NIH); UC4DK117009 (NIH)
Record Dates: First submitted 2013-01-10; First posted 2013-01-23 (Estimated); Results first posted 2024-06-06 (Actual); Last update posted 2024-06-06 (Actual); Status verified 2023-07

CONDITIONS: Abnormal Glucose Tolerance; Type 1 Diabetes
Keywords: prevention of type 1 diabetes; prevention of abnormal glucose tolerance
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Abatacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- abatacept IV infusion (Experimental): CTLA4-Ig (Abatacept) will be administered as 14 (30 minute) infusions over one year (3 infusions every other week the first month; monthly for the following 11 months)
  Interventions: Drug: CTLA4-Ig (Abatacept)
- Placebo (Placebo Comparator): The placebo arm will receive 14 (30 minute) IV infusions (containing saline) given 3 times (every other week) the first month and monthly for the following 11 months.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CTLA4-Ig (Abatacept) — Given as 30 minute IV infusion
  Other Names: Abatacept
  Arms: abatacept IV infusion
Drug: Placebo — Saline given as 30 minute IV infusion
  Arms: Placebo

SUMMARY:
The study is a 2-arm, multicenter, 1:1 randomized, placebo controlled clinical trial.

All subjects will receive close monitoring for development of AGT or T1DM. Subjects will receive Abatacept or placebo and close monitoring for development of AGT or T1DM. To assess the safety, efficacy, and mode of action of Abatacept to prevent AGT and T1DM.

The primary objective is to determine whether intervention with Abatacept will prevent or delay the development of AGT in at-risk autoantibody positive non-diabetic relatives of patients with T1DM.

Secondary outcomes include: the effect of Abatacept on the incidence of T1DM; analyses of C-peptide and other measures from the OGTT; safety and tolerability; and mechanistic outcomes.

DETAILED DESCRIPTION:
Study Purpose and Rationale:

In this study, relatives who are confirmed to have two or more antibodies, not including mIAA, and normal glucose tolerance will be eligible for randomization to experimental treatment or placebo groups with the aim to determine whether experimental treatment will prevent or delay the occurrence of abnormal glucose tolerance and type 1 diabetes mellitus. Individuals with normal glucose tolerance are earlier in the disease process; that is, have less beta cell destruction than those with abnormal glucose tolerance or frank diabetes, yet will inevitably progress to clinical disease and essentially complete beta cell loss. Treatment at this early stage in a population who will inevitably progress to type 1 diabetes provides the greatest opportunity for a clinically important impact on disease prevention. With abnormal glucose tolerance rather than diabetes as the primary endpoint, study participants, regulators, funders, and investigators will be able to determine whether the therapy can alter disease progression.

Therefore, the rationale for this study is that individuals with immunologic markers of T1DM and normal glucose tolerance will inevitably develop clinical T1DM. Prior to development of clinical T1DM they will progress from normal glucose tolerance to abnormal glucose tolerance; and abnormal glucose tolerance results in clinical T1DM within 5 years in almost 80% of subjects. They have a condition that differs from overt diabetes only in the duration of the autoimmune process that results in beta cell destruction. Intervention early in the course of disease may be more effective than intervention in those with abnormal glucose tolerance or clinical T1DM.

Description of Treatment Groups

Subjects will be randomized to receive either Abatacept or placebo infusions along with close monitoring for abnormal glucose tolerance or diabetes. The infusions will be conducted at approved TrialNet clinical sites with appropriate facilities. All blood and serum samples for the primary and secondary outcome determinations will be sent to the Core Laboratories for analysis. Clinical laboratory studies may be done at the local sites.

Participants will be randomly assigned in a 1:1 ratio (within the two strata defined by age at enrollment: <18 and 18 or older) to the following 2 groups:

* to receive Abatacept (intravenous infusion at 0, 2, and 4 weeks following randomization, and then every 28+/-7 days) thereafter for a total of 14 doses. Close monitoring for diabetes development through the duration of study.
* to receive placebo intravenous infusion at 0, 2, and 4 weeks following randomization and then every 28+/- 7 days thereafter for a total of 14 doses. Close monitoring for diabetes development through the duration of study.

Treatment Assignment

After participants sign the consent form, complete the screening visit(s), and meet all of the inclusion criteria and none of the exclusion criteria, participants will be randomized to receive either Abatacept and close monitoring or placebo with close monitoring.

Participants will be randomized in equal allocations to each group. The randomization method will be stratified by TrialNet study site and whether the participant is less than 18 years of age or 18 years and older. This approach ensures that study site will not be a potential confounder. The TNCC will generate the randomization numbers and tables.

Study Assessments

During the course of the study, participants will frequently undergo assessments of their glucose tolerance status, insulin production, immunologic status, and overall health and well-being.

Samples will be drawn for storage in the National Institute for Diabetes and Digestive and Kidney Disease (NIDDK) Repository and at TrialNet Laboratory Sites for future analysis related to T1DM.

Study Duration

The study has been designed to provide 80% power to detect a 40% risk reduction in the occurrence of abnormal glucose tolerance using a two-sided test at the 0.05 level after six years of study duration. A total of approximately 206 patients will be allocated in a 1:1 ratio to the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Participant in TrialNet Natural History/Pathway to Prevention Study and thus, a relative of a proband with T1DM.
* Between the ages of 1-45 years at the time of enrollment in TN01 and age ≥ 6 at time of randomization in this trial.
* Willing to provide Informed Consent or have a parent or legal guardian provide informed consent if the subject is <18 years of age.
* Normal glucose tolerance by OGTT confirmed within 7 weeks (no more than 52 days) of baseline (visit 0). If previous abnormal glucose tolerance, has had two consecutive OGTTs with normal glucose tolerance.

  1. Fasting plasma glucose < 110 mg/dL (6.1 mmol/L), and
  2. 2 hour plasma glucose <140 mg/dL (7.8 mmol/L), and
  3. 30, 60, or 90 minute value on OGTT< 200mg/dL (11.1 mmol/L)
* At least two diabetes-related autoantibodies confirmed to be present on two occasions, not including mIAA. Confirmation of 2 positive autoantibodies must occur within the six months prior to randomization, but the confirmation does not have to involve the same 2 autoantibodies.
* Weight ≥ 20 kg at Baseline Visit.
* If a female participant with reproductive potential, willing to avoid pregnancy and undergo pregnancy testing prior to each infusion.
* At least three months from date of last live immunization.
* Willing to forgo live vaccines while receiving treatment on study and for three months following last study drug administration.

Exclusion Criteria:

* Abnormal Glucose Tolerance or Diabetes

  1. Fasting plasma glucose ≥ 110 mg/dL (6.1 mmol/L), or
  2. 2 hour plasma glucose ≥ 140 mg/dL (7.8 mmol/L), or
  3. 30, 60, 90 minute plasma glucose during OGTT ≥ 200 mg/dL (11.1 mmol/L)
* Insulin autoantibodies (mIAA).
* Are immunodeficient or have clinically significant chronic lymphopenia.
* Have an active infection at time of randomization.
* Have a positive PPD test result or history of previously treated TB, or positive interferon-gamma release assay (IGRA) test.
* Be currently pregnant or lactating, or anticipate getting pregnant within 3 months of the last study drug administration.
* Use of medications known to influence glucose tolerance.
* Require use of other immunosuppressive agents.
* Have serologic evidence of current or past HIV, Hepatitis B (positive for Hepatitis B core antibody or surface antigen), or Hepatitis C infection.
* Have serological evidence of current CMV infection.
* Have evidence of active EBV infection.
* Have any complicating medical issues or abnormal clinical laboratory results that interfere with study conduct or cause increased risk. These include pre-existing cardiac disease, COPD, neurological, or blood count abnormalities (such as lymphopenia, leukopenia, or thrombocytopenia).

Ages: 6 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 212 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2021-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla J Greenbaum, MD, Study Chair — Type 1 Diabetes TrialNet
Locations (17):
- United States (16):
  - University of California - San Francisco, San Francisco, California
  - Stanford University Medical Center, Stanford, California
  - Barbara Davis Center for Childhood Diabetes, University of Colorado, Denver, Colorado
  - Yale Medical School, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of Chicago, Chicago, Illinois
  - Indiana University-Riley Hospital for Children, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - Columbia University, New York, New York
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Vanderbilt University, Nashville, Tennessee
  - University of Texas Medical Center at Dallas, Dallas, Texas
  - Baylor College of Medicine, Houston, Texas
  - Benaroya Research Institute at Virginia Mason, Seattle, Washington
- The Hospital for Sick Children, Toronto, Ontario, Canada

REFERENCES:
- [Background] Orban T, Bundy B, Becker DJ, DiMeglio LA, Gitelman SE, Goland R, Gottlieb PA, Greenbaum CJ, Marks JB, Monzavi R, Moran A, Raskin P, Rodriguez H, Russell WE, Schatz D, Wherrett D, Wilson DM, Krischer JP, Skyler JS; Type 1 Diabetes TrialNet Abatacept Study Group. Co-stimulation modulation with abatacept in patients with recent-onset type 1 diabetes: a randomised, double-blind, placebo-controlled trial. Lancet. 2011 Jul 30;378(9789):412-9. doi: 10.1016/S0140-6736(11)60886-6. Epub 2011 Jun 28. PMID 21719096
- [Derived] Leung SS, Borg DJ, McCarthy DA, Boursalian TE, Cracraft J, Zhuang A, Fotheringham AK, Flemming N, Watkins T, Miles JJ, Groop PH, Scheijen JL, Schalkwijk CG, Steptoe RJ, Radford KJ, Knip M, Forbes JM. Soluble RAGE Prevents Type 1 Diabetes Expanding Functional Regulatory T Cells. Diabetes. 2022 Sep 1;71(9):1994-2008. doi: 10.2337/db22-0177. PMID 35713929
- See also: TrialNet — http://www.diabetestrialnet.org

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Abatacept IV Infusion | Placebo
Started | 101 | 111
Completed | 99 | 108
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Abatacept IV Infusion | Placebo | Total
Number analyzed (Participants) | 101 | 111 | 212
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 16.3 [11.9 to 27.5] | 14.9 [11.4 to 22.0] | 15.6 [11.6 to 23.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 57 | 107
  Male | 51 | 54 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 10 | 21
  Not Hispanic or Latino | 84 | 98 | 182
  Unknown or Not Reported | 6 | 3 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 2
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 91 | 102 | 193
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 6 | 5 | 11
Relationship to person with type 1 diabetes [Count of Participants; unit: Participants]
  Sibling(s) | 53 | 56 | 109
  Identical twin | 1 | 2 | 3
  Offspring | 21 | 14 | 35
  Parent(s) | 14 | 23 | 37
  Sibling and another first degree relative | 6 | 9 | 15
  Second degree relative | 4 | 6 | 10
  Third degree relative | 2 | 1 | 3
Autoantibodies positive [Count of Participants; unit: Participants]
  Anti-GAD65 harmonized | 94 | 104 | 198
  Micro insulin | 4 | 2 | 6
  Anti-IA-2 harmonized | 49 | 61 | 110
  Autoantibodies (ICA) | 76 | 79 | 155
  Anti-ZnT8 | 47 | 65 | 112
Autoantibodies titer [Median (Inter-Quartile Range); unit: titers]
  GADA | 317 [91 to 683] | 375 [100 to 707] | 335 [93.8 to 694]
  Micro insulin | 0.002 [0.001 to 0.003] | 0.002 [0.001 to 0.004] | 0.002 [0.001 to 0.003]
  Anti-IA-2 harmonized | 2 [0 to 225] | 23 [0 to 186] | 9 [0 to 202]
  Autoantibodies (ICA) | 40 [10 to 160] | 40 [5 to 160] | 40 [5 to 160]
  Anti-ZnT8 | 0.013 [0.001 to 0.168] | 0.041 [0.002 to 0.170] | 0.027 [0.001 to 0.169]
Glycated hemoglobin level [Median (Inter-Quartile Range); unit: percentage of glycated hemoglobin] | 5.1 [4.9 to 5.3] | 5.1 [4.9 to 5.25] | 5.1 [4.9 to 5.3]
Body Mass Index (BMI) [Median (Inter-Quartile Range); unit: kg/m^2] | 22.7 [18.5 to 27.3] | 21.6 [17.6 to 25.6] | 22.1 [17.8 to 26.3]
Body Mass Index (BMI) Z-score [Median (Inter-Quartile Range); unit: Z-score] — The BMI Z-score indicates the number of standard deviations away from the mean. A Z-score of 0 is equal to the mean of a reference population (i.e., healthy, age and sex-matched children). Negative numbers indicate values lower than the reference population and positive numbers indicate values higher than the reference population
  Z-score | 0.668 [-0.129 to 1.29] | 0.582 [-0.213 to 1.25] | 0.623 [0.162 to 1.27]
HLA alleles present [Count of Participants; unit: Participants]
  DR3 | 47 | 60 | 107
  DR4 | 60 | 63 | 123
  Missing | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Time From Randomization to Confirmed Abnormal Glucose Tolerance Test
Description: Measured by Oral Glucose Tolerance Test (OGTT):
  Abnormal Glucose Tolerance is primary endpoint and defined as:
  1. Fasting plasma glucose ≥ 110 mg/dL (6.1 mmol/L) and < 126 mg/dL (7 mmol/L), or
  2. 2 hour plasma glucose ≥ 140 mg/dL (7.8 mmol/L) and < 200 (11.1 mmol/L), or
  3. 30, 60, 90 minute plasma glucose during OGTT ≥ 200 mg/dL (11.1 mmol/L)
Time Frame: 96 months
Population: Relatives of patients with type 1 diabetes who did not have diabetes but were at high risk for development of clinical disease.
Measure: Median (Inter-Quartile Range); unit: months
Arm/Group | Abatacept IV Infusion | Placebo
Number analyzed (Participants) | 101 | 111
months | 89.2 [41.1 to NA] — upper quartile range is unknown as it has not been reached | 71.6 [23.7 to NA] — upper quartile range is unknown as it has not been reached

2. Secondary Outcome: Change in C-peptide Concentration to Oral Glucose Tolerance Test (OGTT)
Description: To Determine whether treatment with Abatacept is superior to placebo with respect to C-peptide response to oral glucose tolerance
Time Frame: 0 time to 30 months
Measure: Mean (Inter-Quartile Range); unit: nmol/L
Arm/Group | Abatacept IV Infusion | Placebo
Number analyzed (Participants) | 101 | 111
nmol/L | 2.16 [1.61 to 2.50] | 2.07 [1.51 to 2.74]

ADVERSE EVENTS:
Time Frame: Baseline Visit through study endpoint, up to 6 years
Description: CTCAE; Adverse events were analyzed and published based on organ system class without regard to the specific Adverse Event Term.
Arm/Group | Abatacept IV Infusion | Placebo
All-Cause Mortality (participants affected / at risk) | 0/101 | 0/111
Serious Adverse Events (participants affected / at risk) | 2/101 | 3/111
Other Adverse Events (participants affected / at risk) | 63/101 | 77/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept IV Infusion (N=101) | Placebo (N=111)
Surgical and medical procedures - Other, specify (Surgical and medical procedures) | 0 | 1
Stroke (Nervous system disorders) | 0 | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Appendicitis (Infections and infestations) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Abatacept IV Infusion (N=101) | Placebo (N=111)
Infections and infestations (Infections and infestations) | 38 | 45
Gastrointestinal Disorders (Gastrointestinal disorders) | 22 | 29
Musculoskeletal and Connective Tissue (Musculoskeletal and connective tissue disorders) | 19 | 15
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 16 | 15
General disorders and administration site (General disorders) | 14 | 20
Skin and subcutaneous tissue disorders (Skin and subcutaneous tissue disorders) | 17 | 10
Nervous system disorders (Nervous system disorders) | 13 | 8
Injury, poisoning and procedural (Injury, poisoning and procedural complications) | 15 | 8
Psychiatric disorders (Psychiatric disorders) | 7 | 9
Surgical and medical procedures (Surgical and medical procedures) | 9 | 9
Investigations (Investigations) | 3 | 10
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 5 | 4
Eye disorders (Eye disorders) | 5 | 4
Reproductive system and breast disorders (Reproductive system and breast disorders) | 3 | 3
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 3 | 7
Cardiac disorders (Cardiac disorders) | 3 | 3
Vascular disorders (Vascular disorders) | 2 | 4
Endocrine disorders (Endocrine disorders) | 3 | 2
Pregnancy, puerperium and perinatal (Pregnancy, puerperium and perinatal conditions) | 2 | 0
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 4 | 2
Immune system disorders (Immune system disorders) | 2 | 3
Renal and urinary disorders (Renal and urinary disorders) | 3 | 1
Ear and labyrinth disorders (Ear and labyrinth disorders) | 2 | 2
Hepatobiliary disorders (Hepatobiliary disorders) | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-06-29): https://cdn.clinicaltrials.gov/large-docs/07/NCT01773707/Prot_000.pdf
  • Statistical Analysis Plan (2021-09-09): https://cdn.clinicaltrials.gov/large-docs/07/NCT01773707/SAP_001.pdf